CLINICAL TRIAL: NCT05149196
Title: Impact of Goal-directed Hemodynamic Management on Occurrence of Acute and Persistent Kidney Injury After Radical Nephrectomy or Nephroureterectomy: A Randomized Controlled Trial
Brief Title: Goal-directed Hemodynamic Management and Kidney Injury After Radical Nephrectomy or Nephroureterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-417
Record Dates: First submitted 2021-11-22; First posted 2021-12-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Nephrectomy; Nephroureterectomy; Hemodynamic Management; Acute Kidney Injury; Chronic Kidney Diseases
Keywords: Nephrectomy; Nephroureterectomy; Hemodynamic Management; Acute Kidney Injury; Chronic Kidney Diseases
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted blood pressure management (Experimental): During anesthesia, hemodynamic managements include active hydration (>10 ml/kg/h), use of inotropes (dobutamine), and forced diuresis; the targets are to maintain pulse pressure variation <9%, mean arterial pressure ≥85 mmHg, and urine output >200 ml/h (3ml/kg/h).
  During the first 48 hours after surgery, systolic blood pressure is maintained ≥110 mmHg or within 20% of baseline by delaying antihypertensive resumption, providing fluid challenge, and/or vasoactive infusion.
  Interventions: Other: Targeted hemodynamic management
- Routine care (Active Comparator): During anesthesia, hemodynamic managements are conducted according to routine practice and usually include fluids infusion at a rate of 6-8 ml/kg/h without inotropics; the targets are to maintain mean arterial pressure ≥60 mmHg and urine output >0.5 ml/kg/h.
  During the first 48 hours after surgery, hemodynamic management is performed according to routine practice.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Targeted hemodynamic management — During anesthesia, hemodynamic managements include active hydration (>10 ml/kg/h), use of inotropes (dobutamine), and forced diuresis; the targets are to maintain pulse pressure variation <9%, mean arterial pressure ≥85 mmHg, and urine output >200 ml/h (3ml/kg/h).
  During the first 48 hours after surgery, systolic blood pressure is maintained ≥110 mmHg or within 20% of baseline by delaying antihypertensive resumption, providing fluid challenge, and/or vasoactive infusion.
  Arms: Targeted blood pressure management
Other: Routine care — During anesthesia, hemodynamic managements are conducted according to routine practice and usually include fluid infusion at a rate of 6-8 ml/kg/h without inotropics; the targets are to maintain mean arterial pressure ≥60 mmHg and urine output >0.5 ml/kg/h.
  During the first 48 hours after surgery, hemodynamic management is performed according to routine practice.
  Arms: Routine care

SUMMARY:
Radical nephrectomy and nephroureterectomy are common operations for the treatment of renal cell carcinoma and upper tract urothelial carcinoma, respectively. However, acute kidney injury frequently occurs after surgery. And the occurrence of acute kidney injury is associated with an increased risk of chronic kidney disease. Intraoperative hypotension is identified as an important risk factor of postoperative acute kidney injury. Preliminary studies showed that goal-directed hemodynamic management may reduce kidney injury after surgery but requires further demonstration. We hypothesized that goal-directed hemodynamic management combining hydration, inotropes, and forced diuresis to maintain pulse pressure variation <9%, mean arterial pressure ≥85 mmHg, and urine flow rate >200 ml/h (3 ml/kg/h) may reduce the incidence of acute kidney injury and improve long-term renal outcome after radical nephrectomy or nephroureterectomy. The purpose of this study is to investigate the effect of goal-directed hemodynamic management on the occurrence of acute and persistent kidney injury in patients following radical nephrectomy and nephroureterectomy.

DETAILED DESCRIPTION:
Renal cancer accounts for 20.3% of urinary system tumors, and the incidence is still increasing. Surgical resection is the main treatment of renal cancer; radical nephrectomy is the standard operation for renal cancer of stage T2 or above. For upper tract urothelial carcinoma (UTUC) which includes renal pelvis cancer and ureteral cancer, radical nephroureterectomy is the gold standard treatment. Both procedures involve the removal of one kidney. Acute kidney injury (AKI) is a common complication after radical nephrectomy and nephroureterectomy, with reported incidence from 53.9% to 72.7%. AKI is associated with the development of chronic kidney disease (CKD) and is an independent risk factor of new onset CKD in patients without underlying kidney disease. A meta-analysis showed that, at one year after surgery, patients with AKI had a 2.7-fold increased risk of new onset or progression of CKD and a 4.8-fold increased risk of end-stage renal disease. Moreover, even mild AKI is associated with renal insufficiency at 1 to 2 years after surgery.

Taking active measures to reduce the incidence of AKI may improve long-term renal function after radical nephrectomy and nephroureterectomy. Many clinical studies show that intraoperative hypotension is an important risk factor of postoperative kidney injury. For example, a study found that intraoperative mean arterial pressure (MAP) <65 mmHg or a decrease of more than 20% from baseline was associated with an increased risk of postoperative AKI; the risk of AKI increased alone with prolonged duration of hypotension. However, recent randomized controlled trials showed inconsistent results regarding the effect of tight blood pressure management strategy on kidney outcome. Relevant studies indicated that hydration with forced diuresis and inotropes to maintain cardiac output and blood pressure might improve renal outcome.

In a previous pilot trial of the authors, goal-directed hemodynamic management combining hydration and inotropics reduced the incidence of AKI by about 40% in patients following partial nephrectomy. However, the difference was not statistically significant due to insufficient sample size. The purpose of this trial is to investigate whether goal-directed intraoperative hemodynamic management combining hydration, inotropics, and forced diuresis can reduce the occurrence of acute and persistent kidney injury in patients undergoing radical nephrectomy and nephroureterectomy.

ELIGIBILITY:
Inclusion criteria:

1. Age of 18 years or older;
2. Scheduled to undergo unilateral radical nephrectomy for renal cancer or unilateral radical nephroureterectomy for upper tract urothelial carcinoma.

Exclusion criteria

1. Diagnosed with chronic kidney disease stage 4 or stage 5 (GFR<30 ml/min/1.73m2) before surgery;
2. Uncontrolled severe hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg);
3. Combined with cardiovascular diseases with Revised Cardiac Risk Index (RCRI) >1 or metabolic equivalents (METs) <4;
4. Unable to communicate due to severe dementia, language barrier, or end-stage disease before surgery;
5. Other conditions that are considered unsuitable for inclusion (specific reasons should be indicated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1724 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2032-12-30 (Estimated); Study Completion 2034-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury (early primary outcome) | Up to 7 days after surgery
  Acute kidney injury is diagnosed and classified according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria. Acute kidney injury of stage 1 or above is defined as occurrence of acute kidney injury.
Time to new-onset or progression of chronic kidney disease (CKD) (long-term primary outcome). | Up to 2 years after surgery
  New-onset CKD is defined as a decrease of glomerular filtration rate to <60 ml/min/1.73 m2 and persists for more than 3 months. Progression of CKD is defined as a decrease of glomerular filtration rate of 40% or more from baseline and persists for more than 3 months.

SECONDARY OUTCOMES:
Incidence of myocardial injury after noncardiac surgery (MINS) within 7 days after surgery | Up to 7 days after surgery
  MINS is diagnosed according to the Fourth Universal Definition of Myocardial Infarction (2018).
Incidence of delirium within 7 days after surgery | Up to 7 days after surgery
  Delirium is assessed twice daily with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or the 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM).
Incidence of surgical site infection within 30 days after surgery | Up to 30 days after surgery
  Surgical site infection is diagnosed according to predefined definition.
Incidence of CKD within 3 months after surgery | Up to 3 months after surgery
  Included new-onset or progression of CKD. New-onset CKD is defined as a decrease of glomerular filtration rate to <60 ml/min/1.73 m2 and persists for more than 3 months. Progression of CKD is defined as a decrease of glomerular filtration rate of 40% or more from baseline and persists for more than 3 months.
Proportion of various grades of CKD at different timepoints | Up to 2 years after surgery
  CKD is diagnosed and classified according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria.
Event-free survival | Up to 2 years after surgery
  Time interval from the end of surgery to new-onset or progression of CKD, serious events (required hospitalization or reoperation), or all-cause death, which ever come first. New-onset CKD is defined as a decrease of glomerular filtration rate to <60 ml/min/1.73 m2 and persists for more than 3 months. Progression of CKD is defined as a decrease of glomerular filtration rate of 40% or more from baseline and persists for more than 3 months.

OTHER OUTCOMES:
AKI stage within 7 days after surgery | Up to 7 days after surgery
  Acute kidney injury is diagnosed and classified according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria.
Proportion of patients admitted in intensive care unit after surgery | Up to 30 days after surgery
  Proportion of patients admitted in intensive care unit after surgery.
Incidence of other major postoperative complications | Up to 30 days after surgery
  Major postoperative complications are defined as new-onset medical conditions that are harmful to patients' recovery and required therapeutic intervention, i.e., grade 2 or higher on the Clavien-Dindo classification.
Length of hospital stay after surgery | Up to 30 days after surgery
  Length of hospital stay after surgery
Prevalence of neurocognitive disorder at 6 months and 1 year after surgery | At 6 months and 1 year after surgery
  Neurocognitive disorder is defined as a decrease of neurocognitive function score of 1 standard deviation (SD) or more from baseline. Neurocognitive function is assessed with the Montreal Cognitive Assessment-telephone version (T-MoCA; score ranges from 0 to 22, with higher score indicating better cognitive function).
Quality of life at 6 months and 1 year after surgery | At 6 months and 1 year after surgery
  Quality of life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF), a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.
Overall survival time | Up to 2 years after surgery
  Time interval from the end of surgery to all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Klatte T, Rossi SH, Stewart GD. Prognostic factors and prognostic models for renal cell carcinoma: a literature review. World J Urol. 2018 Dec;36(12):1943-1952. doi: 10.1007/s00345-018-2309-4. Epub 2018 Apr 30. PMID 29713755
- [Background] Cho A, Lee JE, Kwon GY, Huh W, Lee HM, Kim YG, Kim DJ, Oh HY, Choi HY. Post-operative acute kidney injury in patients with renal cell carcinoma is a potent risk factor for new-onset chronic kidney disease after radical nephrectomy. Nephrol Dial Transplant. 2011 Nov;26(11):3496-501. doi: 10.1093/ndt/gfr094. Epub 2011 Mar 15. PMID 21406544
- [Background] Garofalo C, Liberti ME, Russo D, Russo L, Fuiano G, Cianfrone P, Conte G, De Nicola L, Minutolo R, Borrelli S. Effect of post-nephrectomy acute kidney injury on renal outcome: a retrospective long-term study. World J Urol. 2018 Jan;36(1):59-63. doi: 10.1007/s00345-017-2104-7. Epub 2017 Oct 23. PMID 29063267
- [Background] Shin S, Han Y, Park H, Chung YS, Ahn H, Kim CS, Cho YP, Kwon TW. Risk factors for acute kidney injury after radical nephrectomy and inferior vena cava thrombectomy for renal cell carcinoma. J Vasc Surg. 2013 Oct;58(4):1021-7. doi: 10.1016/j.jvs.2013.02.247. Epub 2013 Apr 13. PMID 23591189
- [Background] Chawla LS, Eggers PW, Star RA, Kimmel PL. Acute kidney injury and chronic kidney disease as interconnected syndromes. N Engl J Med. 2014 Jul 3;371(1):58-66. doi: 10.1056/NEJMra1214243. No abstract available. PMID 24988558
- [Background] See EJ, Jayasinghe K, Glassford N, Bailey M, Johnson DW, Polkinghorne KR, Toussaint ND, Bellomo R. Long-term risk of adverse outcomes after acute kidney injury: a systematic review and meta-analysis of cohort studies using consensus definitions of exposure. Kidney Int. 2019 Jan;95(1):160-172. doi: 10.1016/j.kint.2018.08.036. Epub 2018 Nov 23. PMID 30473140
- [Background] Turan A, Cohen B, Adegboye J, Makarova N, Liu L, Mascha EJ, Qiu Y, Irefin S, Wakefield BJ, Ruetzler K, Sessler DI. Mild Acute Kidney Injury after Noncardiac Surgery Is Associated with Long-term Renal Dysfunction: A Retrospective Cohort Study. Anesthesiology. 2020 May;132(5):1053-1061. doi: 10.1097/ALN.0000000000003109. PMID 31929326
- [Background] Kim WH, Shin KW, Ji SH, Jang YE, Lee JH, Jeong CW, Kwak C, Lim YJ. Robust Association between Acute Kidney Injury after Radical Nephrectomy and Long-term Renal Function. J Clin Med. 2020 Feb 25;9(3):619. doi: 10.3390/jcm9030619. PMID 32106477
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Shin CH, Long DR, McLean D, Grabitz SD, Ladha K, Timm FP, Thevathasan T, Pieretti A, Ferrone C, Hoeft A, Scheeren TWL, Thompson BT, Kurth T, Eikermann M. Effects of Intraoperative Fluid Management on Postoperative Outcomes: A Hospital Registry Study. Ann Surg. 2018 Jun;267(6):1084-1092. doi: 10.1097/SLA.0000000000002220. PMID 28288059
- [Background] Myles PS, McIlroy DR, Bellomo R, Wallace S. Importance of intraoperative oliguria during major abdominal surgery: findings of the Restrictive versus Liberal Fluid Therapy in Major Abdominal Surgery trial. Br J Anaesth. 2019 Jun;122(6):726-733. doi: 10.1016/j.bja.2019.01.010. Epub 2019 Feb 16. PMID 30916001
- [Background] Giglio M, Dalfino L, Puntillo F, Brienza N. Hemodynamic goal-directed therapy and postoperative kidney injury: an updated meta-analysis with trial sequential analysis. Crit Care. 2019 Jun 26;23(1):232. doi: 10.1186/s13054-019-2516-4. PMID 31242941
- [Background] Kellum JA, Ronco C, Mehta RL. Fluid management in acute kidney injury. Int J Artif Organs. 2008 Feb;31(2):94-5. doi: 10.1177/039139880803100203. No abstract available. PMID 18311726
- [Background] Wu QF, Kong H, Xu ZZ, Li HJ, Mu DL, Wang DX. Impact of goal-directed hemodynamic management on the incidence of acute kidney injury in patients undergoing partial nephrectomy: a pilot randomized controlled trial. BMC Anesthesiol. 2021 Mar 3;21(1):67. doi: 10.1186/s12871-021-01288-8. PMID 33658007
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Ficarra V, Novara G, Secco S, Macchi V, Porzionato A, De Caro R, Artibani W. Preoperative aspects and dimensions used for an anatomical (PADUA) classification of renal tumours in patients who are candidates for nephron-sparing surgery. Eur Urol. 2009 Nov;56(5):786-93. doi: 10.1016/j.eururo.2009.07.040. Epub 2009 Aug 4. PMID 19665284
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Pancaro C, Shah N, Pasma W, Saager L, Cassidy R, van Klei W, Kooij F, Vittali D, Hollmann MW, Kheterpal S, Lirk P. Risk of Major Complications After Perioperative Norepinephrine Infusion Through Peripheral Intravenous Lines in a Multicenter Study. Anesth Analg. 2020 Oct;131(4):1060-1065. doi: 10.1213/ANE.0000000000004445. PMID 32925324
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Chiu C, Fong N, Lazzareschi D, Mavrothalassitis O, Kothari R, Chen LL, Pirracchio R, Kheterpal S, Domino KB, Mathis M, Legrand M. Fluids, vasopressors, and acute kidney injury after major abdominal surgery between 2015 and 2019: a multicentre retrospective analysis. Br J Anaesth. 2022 Sep;129(3):317-326. doi: 10.1016/j.bja.2022.05.002. Epub 2022 Jun 8. PMID 35688657
- [Background] Briguori C, D'Amore C, De Micco F, Signore N, Esposito G, Visconti G, Airoldi F, Signoriello G, Focaccio A. Left Ventricular End-Diastolic Pressure Versus Urine Flow Rate-Guided Hydration in Preventing Contrast-Associated Acute Kidney Injury. JACC Cardiovasc Interv. 2020 Sep 14;13(17):2065-2074. doi: 10.1016/j.jcin.2020.04.051. PMID 32912462
- [Background] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Reduction in acute kidney injury post cardiac surgery using balanced forced diuresis: a randomized, controlled trial. Eur J Cardiothorac Surg. 2021 Apr 13;59(3):562-569. doi: 10.1093/ejcts/ezaa395. PMID 33236105
- [Background] Wu X, Jiang Z, Ying J, Han Y, Chen Z. Optimal blood pressure decreases acute kidney injury after gastrointestinal surgery in elderly hypertensive patients: A randomized study: Optimal blood pressure reduces acute kidney injury. J Clin Anesth. 2017 Dec;43:77-83. doi: 10.1016/j.jclinane.2017.09.004. Epub 2017 Oct 19. PMID 29055803
- [Background] Wanner PM, Wulff DU, Djurdjevic M, Korte W, Schnider TW, Filipovic M. Targeting Higher Intraoperative Blood Pressures Does Not Reduce Adverse Cardiovascular Events Following Noncardiac Surgery. J Am Coll Cardiol. 2021 Nov 2;78(18):1753-1764. doi: 10.1016/j.jacc.2021.08.048. PMID 34711333
- [Background] Marcucci M, Painter TW, Conen D, Lomivorotov V, Sessler DI, Chan MTV, Borges FK, Leslie K, Duceppe E, Martinez-Zapata MJ, Wang CY, Xavier D, Ofori SN, Wang MK, Efremov S, Landoni G, Kleinlugtenbelt YV, Szczeklik W, Schmartz D, Garg AX, Short TG, Wittmann M, Meyhoff CS, Amir M, Torres D, Patel A, Ruetzler K, Parlow JL, Tandon V, Fleischmann E, Polanczyk CA, Lamy A, Jayaram R, Astrakov SV, Wu WKK, Cheong CC, Ayad S, Kirov M, de Nadal M, Likhvantsev VV, Paniagua P, Aguado HJ, Maheshwari K, Whitlock RP, McGillion MH, Vincent J, Copland I, Balasubramanian K, Biccard BM, Srinathan S, Ismoilov S, Pettit S, Stillo D, Kurz A, Belley-Cote EP, Spence J, McIntyre WF, Bangdiwala SI, Guyatt G, Yusuf S, Devereaux PJ; POISE-3 Trial Investigators and Study Groups. Hypotension-Avoidance Versus Hypertension-Avoidance Strategies in Noncardiac Surgery : An International Randomized Controlled Trial. Ann Intern Med. 2023 May;176(5):605-614. doi: 10.7326/M22-3157. Epub 2023 Apr 25. PMID 37094336
- [Background] Saugel B, Fletcher N, Gan TJ, Grocott MPW, Myles PS, Sessler DI; PeriOperative Quality Initiative XI (POQI XI) Workgroup Members. PeriOperative Quality Initiative (POQI) international consensus statement on perioperative arterial pressure management. Br J Anaesth. 2024 Aug;133(2):264-276. doi: 10.1016/j.bja.2024.04.046. Epub 2024 Jun 4. PMID 38839472
- [Background] Dudinec JV, Ortiz-Melo DI, Lipkin ME, Abern MR, Shah AM, Inman BA. Advanced chronic kidney disease; A comparison between nephroureterectomy and nephron-sparing surgery for upper tract urothelial carcinoma. Urol Oncol. 2023 Jun;41(6):295.e19-295.e25. doi: 10.1016/j.urolonc.2022.11.020. Epub 2022 Dec 14. PMID 36526526
- [Background] Tafuri A, Marchioni M, Cerrato C, Mari A, Tellini R, Odorizzi K, Veccia A, Amparore D, Shakir A, Carbonara U, Panunzio A, Trovato F, Catellani M, Janello LMI, Bianchi L, Novara G, Dal Moro F, Schiavina R, De Lorenzis E, Parma P, Cimino S, De Cobelli O, Maiorino F, Bove P, Crocerossa F, Cantiello F, D'Andrea D, Di Cosmo F, Porpiglia F, Ditonno P, Montanari E, Soria F, Gontero P, Liguori G, Trombetta C, Mantica G, Borghesi M, Terrone C, Del Giudice F, Sciarra A, Galosi A, Moschini M, Shariat SF, Di Nicola M, Minervini A, Ferro M, Cerruto MA, Schips L, Pagliarulo V, Antonelli A. Changes in renal function after nephroureterectomy for upper urinary tract carcinoma: analysis of a large multicenter cohort (Radical Nephroureterectomy Outcomes (RaNeO) Research Consortium). World J Urol. 2022 Nov;40(11):2771-2779. doi: 10.1007/s00345-022-04156-3. Epub 2022 Oct 6. PMID 36203101
- [Background] Tafuri A, Odorizzi K, Di Filippo G, Cerrato C, Fassio G, Serafin E, Princiotta A, D'Aietti D, Gozzo A, Porcaro AB, Brunelli M, Cerruto MA, Antonelli A. Acute kidney injury strongly influences renal function after radical nephroureterectomy for upper tract urothelial carcinoma: A single-centre experience. Arch Ital Urol Androl. 2021 Mar 18;93(1):9-14. doi: 10.4081/aiua.2021.1.9. PMID 33754601